CLINICAL TRIAL: NCT05325073
Title: Erythropoietin Therapy to Induce Regulatory T Cells in Liver Transplant Recipients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Josh Levitsky, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00215838
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplant Rejection
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EPO Arm (Other)
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Erythropoietin

SUMMARY:
The hypothesis of this proof-of-concept study is that EPO increases the frequency, stability and/or function of Tregs in liver transplant recipients. We also hypothesize that EPO will have a greater effect in everolimus vs. tacrolimus treated LTR, thus providing the rationale for a subsequent clinical trial to utilize EPO in combination with everolimus as a more successful pathway toward tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-74 years
* History of liver transplantation > 2 years prior for non-immune causes
* Use of immunosuppressive monotherapy (either tacrolimus or everolimus) for treatment of liver transplantation
* Stable immunosuppression regimen at least 3 months prior to enrollment.
* Ability to provide verbal and written informed consent

Exclusion Criteria:

* • Hgb above average normal value (15.7 g/dL in men, 13.8 g/dL in women); ALT > 2 times upper limit of normal; uncontrolled hypertension with SBP>160 or DBP>100; end-stage renal disease on hemodialysis; history of venous thromboembolism including deep vein thromboses or pulmonary emboli, stroke, heart failure, seizure disorder, significant cardiovascular disease including a history of myocardial infarction, pure red cell aplasia, intolerance or allergy to erythropoietin; Active malignancy (untreated or undergoing therapy); known hypersensitivity to mammalian cell-derived products; known hypersensitivity to human albumin; presence of vascular access; prior recipient of erythropoietin within 12 weeks of the study; and pregnancy

  * Patient unable to provide consent including infants, children, teenagers, prisoners, cognitively impaired adults.
  * Prisoners and other vulnerable populations will also be excluded

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
EPO effects on Treg induction | 12 weeks
  We will use flow cytometry to analyze the phenotype of peripheral blood mononuclear cells (PBMC) collected before and 4 and 12 weeks after EPO administration. Data will be analyzed to extract changes in lymphocyte subset frequencies, including Tregs

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No